CLINICAL TRIAL: NCT02250001
Title: Asunaprevir/Daclatasvir Safety Surveillance in Japanese Patients With Chronic Hepatitis C
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI444-244
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Chronic Hepatitis C
Keywords: HCV
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 48 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment with DCV/ASV: Patients who are beginning to receive the treatment with DCV/ASV under the approved indications, dosage, and administration will be included in this study

SUMMARY:
The primary objective of this study is: To evaluate the real-world safety, specifically the incidence rates of hepatic toxicity, pyrexia, and resistance, of DCV/ASV dual therapy in Japanese patients chronically infected with HCV GT-1.

DETAILED DESCRIPTION:
Time Perspective: Other - For patients who are treated before the contract between Bristol-Myers Kabushiki Kaisha (BMKK) and the treating physician is initiated, patient data will be collected retrospectively after the contract is signed. Data will be collected prospectively for patients who initiate DCV/ASV treatment after the contract is initiated

Patient Registry study - Yes; 48 weeks (Treatment: 24 weeks, Follow up: 24 weeks)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Patients who are initiating DCV and ASV treatment for the first time under the approved indications, dosage, and administration will be included in this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University hospitals, General hospitals, and clinics that have relevant departments, such as Liver Internal medicine, Gastroenterological medicine, Internal medicine, etc, where the surveillance drug is mainly prescribed
Sampling Method: Probability Sample
Enrollment: 2974 (Actual)
Dates: Start 2014-09-30 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
The real-world safety, specifically the incidence rates of hepatic toxicity, pyrexia, and resistance, of Daclatasvir/Asunaprevir (DCV/ASV) dual therapy in Japanese patients chronically infected with Hepatitis C virus Genotype 1 (HCV GT-1) | 28 weeks

SECONDARY OUTCOMES:
Antiviral activity as determined by the proportion of patients with sustained virologic response at 24 weeks post-treatment Sustained virologic response at 24 weeks post-treatment (SVR24) | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Chuo-ku, Tokyo, Japan

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx